CLINICAL TRIAL: NCT02987634
Title: Phase IV Study to Evaluate and Compare the Efficacy of PeriActive Mouthwash to Chlorhexidine 0.12% Rinse With Regards to Managing Post-surgical Inflammation Associated With Dental Implant Surgery
Brief Title: Evaluation and Comparison of Efficacy of PeriActive Mouthwash to Chlorhexidine 0.12% Mouth Rinse
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izun Pharma Ltd (Industry)
Collaborators: Jerusalem Perio Center (Unknown); Herzog Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PORPIS
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Periodontal Diseases
Keywords: gingivitis; dental implant; mouthwash
MeSH Terms: conditions — Periodontal Diseases; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PeriActive mouthwash (Experimental): patient is directed to rinse twice a day for 4 weeks. each rinse is 15 ml of Periactive
  Interventions: Other: PeriActive
- chlorhexidine 0.12% mouthwash (Active Comparator): patient is directed to rinse twice a day for 4 weeks. each rinse is 10 ml of Periactive
  Interventions: Other: PeriActive

INTERVENTIONS:
Other: PeriActive — mouthwash

SUMMARY:
Izun Pharmaceuticals has shown that PeriActive, an oral rinse containing extracts of Sambucus nigra, Echinacea purpurea, and Centella asiatica significantly reduced gingival inflammation in an experimental gingivitis model in a phase II study, as well as in numerous other clinical trials. The product and its individual components were shown to be safe.

Based on these favorable results, Izun is now seeking to demonstrate that a combined anti-bacterial/anti-inflammatory rinse will potentially enhance soft tissue healing and reduce localized inflammation following dental implant surgery equal to, or better than, a chlorhexidine rinse, with fewer side effects.

DETAILED DESCRIPTION:
This is a randomized phase IV controlled trial with two parallel arms: (1) PeriActive rinse and (2) Chlorhexidine 0.12% rinse. Subjects will be randomized to one of two treatment groups at the time of implant surgery. An alternating 1:1 randomization scheme will be used, with the first patient receiving Chlorhexidine, the second patient receiving PeriActive, the third patient receiving Chlorhexidine and so forth.

Implant surgery will require an incision and tissue reflection. Implant(s) will be placed at bone level (+/- 2 mm). The abutment placed will be transgingival at least 2 mm above soft tissue level. Tissues will be sutured with 6-0 ePTFE (Goretex) sutures, as needed. Antibiotics will be prescribed for 7 days following surgery. In addition, at the end of the surgical visit, the patient will be issued two bottles of the assigned rinse which will be used twice each day.

Details of Study Visits Screening/Visit 1 - Day 0 Following signing of informed consent form, adult male and female subjects aged ≥18 years will be screened for study eligibility by assessment of inclusion and exclusion criteria. Screening procedures will include collection of demographic data and medical history. Eligible subjects will then undergo implant surgery, and relevant indices will be measured. Subjects will then be instructed in how to rinse with the relevant oral rinse and be given two bottles for the remainder of the study.

Visits 2 and 3 - 2 and 4 weeks (± 3 days) post-surgery, respectively At visit 2, sutures will be removed and a light curetting of the sites (as needed) will be performed, followed by evaluation for Gingival Index (GI; modified for incision), Plaque Index (PI) and compliance with protocol. At visit 3, only clinical indices and compliance with protocol with be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be adult males or females over the age of 18 years.
2. Subjects must be able and willing to follow study procedures and instructions.
3. Subjects must present with the need for implant surgery that would necessitate surgical incision (flap elevation) and transgingival implant healing cap, be available for follow-up visits and be able to follow rinse protocol instructions.

Exclusion Criteria:

1. Subjects who exhibit gross oral pathology and severe gingival inflammation at the time of surgery at the projected surgical site.
2. Subjects chronically treated (i.e., ≥ two weeks) with anti-inflammatory medications (steroids or nonsteroidal anti-inflammatory drugs) or any other medications known to affect gingival tissue status (e.g., phenytoin, cyclosporine) within one month of the screening examination. Prophylactic use of aspirin ( 81 mg daily) and Plavix when used for cardiovascular indications will be permitted (a note should be inserted into patient's documentation) and any therapeutic treatment modifications will be under the jurisdiction of the treating dentist. All other medications for chronic medical conditions should be initiated at least three months prior to enrollment.
3. Subjects with active infectious diseases such as hepatitis, human immunodeficiency virus (HIV) or tuberculosis
4. Subjects with Types I or II diabetes, thyroid disease or cancer chemotherapy
5. Subjects reporting allergies to the constituents in the rinse
6. Female subjects who report being pregnant or lactating
7. Subjects with clinically significant laboratory results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
GI at buccal margin of implant | 2-4 weeks
GI at margin of flap adjacent to implant | 2-4 weeks

IPD SHARING:
Plan to Share IPD: No
trial results will be published for dentists to see